CLINICAL TRIAL: NCT02512523
Title: A Randomized, Double-blind, Active Control, Parallel Group, Exploratory Phase IV Study to Compare the Effects of Tenelia® or Januvia® on Glucose Variability in add-on to Metformin in Patients With Inadequately Controlled Type2 Diabetes Mellitus in Metformin Only Treatment
Brief Title: Exploratory Study to Compare the Effects of Tenelia® or Januvia® on Glucose Variability in add-on to Metformin (CGMS Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HD_TEN_PH42014
Record Dates: First submitted 2015-07-29; First posted 2015-07-31 (Estimated); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; CGMS; Teneligliptin; Sitagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teneligliptin (Experimental): Film-coated tablet for oral administration Dosage: 20mg/tablet Frequency and duration: 1 tablet/day for 4 weeks
  Interventions: Drug: Teneligliptin
- Sitagliptin (Active Comparator): Film-coated tablet for oral administration Dosage: 100mg/tablet Frequency and duration: 1 tablet/day for 4 weeks
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Teneligliptin
  Arms: Teneligliptin
Drug: Sitagliptin
  Arms: Sitagliptin

SUMMARY:
This is a randomized, double-blind, active control, parallel group, exploratory phase 4 study to compare the effect of teneligliptin versus sitagliptin on glucose variability when added on to metformin in patients with inadequately controlled type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This study will enroll patients with in adequately controlled type 2 diabetes mellitus who have been on metformin (1,000 mg or above) for 8 weeks at least or longer and randomly add teneliglipin (20 mg/day) or sitagliptin (100 mg/day) for 4 weeks. Continuous glucose monitoring will be checked before and after 4-week administration of teneliglipin or sitagliptin together with mixed meal tolerance test (MMTT). Other efficacy and safety parameters will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female aged above (or equal to) 19 years old at screening, inclusive.
2. Patient was diagnosed with type 2 diabetes mellitus at least 3 months prior to screening according to the diagnostic criteria of KDA for at screening
3. Patient has FPG ≤ 270 mg/dl (15.0 mmol/L) at screening
4. Patient who was treated with Metformin (≥1000 mg/day) for at least 8 weeks prior to screening
5. Patient has HbA1c (6.5%≤HbA1c≤9.0%) at screening
6. Patient has adequate renal and hepatic function at screening as defined by the following clinical chemistry results:

   * (male) Serum creatinine <1.5 × upper limit of normal (ULN), (female) Serum creatinine <1.4 × upper limit of normal (ULN),
   * Serum alanine aminotransferase <2.5 × ULN
   * Serum aspartate aminotransferase <2.5 × ULN
7. Both male and female patients and their partners of childbearing potential must agree to use 2 medically accepted methods of contraception (eg, barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], and intrauterine devices) during the course of the study(excluding women who are not of childbearing potential and men who have been sterilized).
8. Male and female patients and their partners who have been surgically sterilized for less than 6 months prior to study entry must agree to use 2 medically accepted methods of contraception as per inclusion criterion 7.
9. Menopausal females must have experienced their last period more than 12 months prior to study entry to be classified as not of childbearing potential.
10. Patient (or legal guardian, if applicable) is informed of the full nature and purpose of the study, including possible risks and side effects, and understand this information, voluntarily signed and dated the written informed consent in compliance with protocol before inclusion in the study

Exclusion Criteria:

1. Patients who have hypersensitivity/allergies to main ingredient of sitagliptin/teneligliptin or any of the excipients of Investigational products(eg. Mannitol).
2. Patient with severe ketosis, diabetic coma or pre coma, Type 1 DM
3. Patient is suffering from any disease, including Type 2 diabetes or its complications that, in the opinion of the Investigator, is sufficiently severe to render the subject unfit, or affect the subject's ability, to participate in the study, for example:

   * Macroangiopathy with symptoms of coronary heart disease or peripheral arterial obstructive disease.
   * Microangiopathy with symptoms of (autonomous) neuropathy with any one or more of the following: gastroparesis
   * Symptoms of poor blood glucose control (polyuria, polydipsia or weight loss)
   * Severe infection, pre or post-operative, severe trauma
4. Patient has a medical history of unstable angina, or heart failure(New York Heart Association class Ⅲ-IV) or any clinically significant ECG abnormalities such as ventricular tachycardia
5. The subject has diastolic blood pressure >100 mmHg and/or systolic blood pressure >180 mmHg at the screening visit
6. Patient who has malignancy at screening or history of any malignancy (except history of no recurrence of malignancy more than 5 years)
7. Female patient whose pregnancy test is negative or who are pregnant, lactating, or are planning to become pregnant during the study
8. Patient is expected to require additional diabetic treatment for his/her Type 2 diabetes or its complications during the study after the screening visit
9. Patient has a history of drug abuse
10. Patient who is under malnutrition, weakness or, in the opinion of the Investigator, patient who drinks on average more than 28 units of alcohol per week (One unit of alcohol equals approximately 250 mL of beer, 125 mL of wine or 40 mL of spirits)
11. Patients taking any of the following concomitant medications:

    * Oral anti-diabetic therapy excluding Metformin within 8 weeks of screening
    * Thiazolidinedione class of drugs within 12 weeks of screening
    * GLP-1 analogues/DPP4 inhibitor class of drugs within 12 weeks of screening(but, following patients will be excluded from the study regardless of treatment duration of previous DPP4 inhibitors: patient who has experienced failure of glucose control with treatment of DPP4 inhibitors or patient who is not expected to have additional good effect of glucose control with administration of IP according to the investigator's opinion)
    * Anti-obesity agent within 12 weeks of screening
    * All kinds of insulin administered within 12 weeks of screening
    * Systemic Corticosteroids or intermittent use of high-dose of steroids(inhaler)
    * Any other investigational drug
12. Patients who have participated in a study with an investigational drug within 12 weeks of Screening or who are currently receiving treatment with any other investigational drug in a study.
13. The presence of any other condition including clinical laboratory test results that leads the investigator to conclude that the patient is inappropriate for inclusion in the clinical study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-08-27 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-26 (Actual)

PRIMARY OUTCOMES:
Mean amplitude of glucose excursion (MAGE) | 4 weeks
  Change in mean amplitude of glucose excursion (MAGE) from baseline at 4 weeks

SECONDARY OUTCOMES:
Standard deviation (SD) | 4 weeks
  Change in standard deviation (SD) from baseline at 4 weeks
Mean blood glucose (MBG) | 4 weeks
  Change in mean blood glucose (MBG) from baseline at 4 weeks
Mixed meal tolerance test (MMTT) | 4 weeks
  Change in Mixed meal tolerance test (MMTT) parameters including glucose, GLP-1, insulin, C-peptide, glucagon, HOMA-IR, HOMA-b from baseline at 4 weeks
Safety (All AE including SAE, hypoglycemia, laboratory tests, vital sign, and physical examination) | 4 weeks
  All AE including SAE, hypoglycemia, laboratory tests, vital sign, and physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Sin Gon Kim, MD, Ph.D, Principal Investigator — Korea University Anam Hospital
Locations (1):
- HANDOK Inc., Seoul, South Korea